CLINICAL TRIAL: NCT00491322
Title: Impact of Vitamin D Deficiency on Insulin Resistance and the Regulation of FGF-23
Brief Title: Vitamin D Deficiency, Insulin Resistance and FGF-23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sherri-Ann M. Burnett-Bowie, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-P-000430/18; K23DK073356 (NIH)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Vitamin D deficiency; Insulin resistance; Diabetes; Diabetes mellitus; FGF-23; FGF23; Phosphate
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Diabetes Mellitus | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergocalciferol group (Experimental): Ergocalciferol 50000 international units once a week for 12 weeks
  Interventions: Dietary Supplement: Ergocalciferol
- Ergocalciferol Placebo group (Placebo Comparator): Matching placebo once a week for 12 weeks
  Interventions: Dietary Supplement: Ergocalciferol placebo

INTERVENTIONS:
Dietary Supplement: Ergocalciferol — Ergocalciferol 50000 international units once a week for 12 weeks
  Arms: Ergocalciferol group
Dietary Supplement: Ergocalciferol placebo — Ergocalciferol placebo once a week for 12 weeks
  Arms: Ergocalciferol Placebo group

SUMMARY:
The purpose of this project is to determine if treating vitamin D deficiency decreases insulin resistance and improves insulin secretion in healthy volunteers. Additionally, this project will investigate if treating vitamin D deficiency affects a new phosphate-regulating hormone called FGF-23.

DETAILED DESCRIPTION:
Vitamin D deficiency or hypovitaminosis D, defined as serum 25 hydroxyvitamin D < or = 20 ng/mL, is prevalent in several populations in the United States, specifically minorities and the elderly. Causes of vitamin D deficiency include lack of exposure to sunlight, malnutrition, and drugs that alter vitamin D metabolism and absorption.

Vitamin D is an essential factor for many organ systems. Data suggest that vitamin D is required for normal insulin secretion by the pancreas. Specifically, animal studies demonstrate that treatment of vitamin D deficiency improves insulin secretion. In humans, there is less consensus about the impact of vitamin D deficiency on insulin resistance. In one study of middle-aged patients with Type 2 diabetes mellitus, no association was seen between serum 25 hydroxyvitamin D levels and a measure of insulin resistance. However, in a larger study of younger glucose tolerant subjects, serum 25 hydroxyvitamin D levels were associated with both insulin secretion and insulin resistance. These data suggest that treatment of vitamin D deficiency may delay or prevent the development of insulin resistance, and thus diabetes mellitus type 2. Repletion of this common vitamin deficiency could therefore have major public health implications for the prevention of diabetes mellitus.

Fibroblast growth factor 23 (FGF-23) is a newly discovered phosphaturic hormone that is regulated by both dietary and serum phosphate. Hormonal regulation of FGF-23, however, is largely unknown. Recent data suggest that vitamin D plays an important role in the regulation of FGF-23. Some groups have shown that inactivation of the vitamin D receptor gene decreases serum FGF-23 levels in mice; administration of 1,25 dihydroxyvitamin D stimulates the transcription of the FGF-23 gene in vitro. Little is known, however, about the regulation of FGF-23 by vitamin D in humans.

Phosphate is critical for bone mineralization, muscle function, signal transduction, and the creation and utilization of energy. Vitamin D deficiency can result in phosphate malabsorption, osteomalacia and increased risk of fractures. Enhanced understanding of the regulation of this new phosphate-regulating hormone, FGF-23, will advance the field of phosphate metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 yrs
* Serum 25-OHD < or = 20 ng/mL
* At least 1 menses in the last 3 months (females) and normal serum testosterone (males)

Exclusion Criteria:

* Significant cardiac, hepatic, oncologic, or psychiatric disease
* History of diabetes mellitus, malabsorption, kidney stones, or recent alcohol excess/abuse (15 drinks per week in the last month)
* Fasting glucose > 126 mg/dl or 2 hour OGTT > 200 mg/dl
* Use of medications known to affect serum phosphate levels including phosphate-binding antacids, sodium etidronate, calcitonin, excessive doses of vitamin D (> 1000 units per day), excessive doses of vitamin A (> 20,000 units/day), calcitriol, growth hormone, or anti-convulsants
* Use of metformin or insulin sensitizing agents
* Serum calcium < 8 or > 11 mg/dL, creatinine > 1.5 mg/dL, or Hgb < 11 gm/dL
* Liver function tests > 2 times the upper limit of normal
* TSH < 0.1 or > 7 uU/mL
* WBC < 2,000 or > 15,000/cmm
* Platelet count < 100,000 or > 500,000/cum
* Hormone replacement therapy or testosterone use
* Urine uhCG positive (females), testosterone < 270 ng/dL (males)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherri-Ann M Burnett-Bowie, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burnett SM, Gunawardene SC, Bringhurst FR, Juppner H, Lee H, Finkelstein JS. Regulation of C-terminal and intact FGF-23 by dietary phosphate in men and women. J Bone Miner Res. 2006 Aug;21(8):1187-96. doi: 10.1359/jbmr.060507. PMID 16869716
- [Background] Burnett-Bowie SM, Mendoza N, Leder BZ. Effects of gonadal steroid withdrawal on serum phosphate and FGF-23 levels in men. Bone. 2007 Apr;40(4):913-8. doi: 10.1016/j.bone.2006.10.016. Epub 2006 Dec 8. PMID 17157573
- [Result] Burnett-Bowie SA, Leder BZ, Henao MP, Baldwin CM, Hayden DL, Finkelstein JS. Randomized trial assessing the effects of ergocalciferol administration on circulating FGF23. Clin J Am Soc Nephrol. 2012 Apr;7(4):624-31. doi: 10.2215/CJN.10030911. Epub 2012 Feb 2. PMID 22300739
- [Derived] Mitchell DM, Leder BZ, Cagliero E, Mendoza N, Henao MP, Hayden DL, Finkelstein JS, Burnett-Bowie SA. Insulin secretion and sensitivity in healthy adults with low vitamin D are not affected by high-dose ergocalciferol administration: a randomized controlled trial. Am J Clin Nutr. 2015 Aug;102(2):385-92. doi: 10.3945/ajcn.115.111682. Epub 2015 Jul 8. PMID 26156733

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 2006-2008. Subjects were healthy volunteers recruited from the community
Groups:
- Placebo Group: Matching placebo once a week for 12 weeks
Period: Overall Study
Arm/Group | Ergocalciferol Group | Placebo Group
Started | 41 | 51
Completed | 40 | 50
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: While 92 subjects were enrolled, 2 subjects, 1 in each group, were withdrawn from the study and their data never analyzed due to pregnancy that prevented initiation of the study drug and 6 week non-compliance with the study medication due to a non-related illness.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol Group | Placebo Group | Total
Number analyzed (Participants) | 40 | 50 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 50 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) | 29 (9) | 28 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 31 | 55
  Male | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 40 | 50 | 90

OUTCOME MEASURES:

1. Primary Outcome: Fibroblast Growth Factor 23 (FGF23) After 12 Weeks of Weekly Ergocalciferol 50000 Units
Description: Fibroblast growth factor 23 (FGF23) is a phosphate and vitamin D regulating hormone.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Ergocalciferol Group: Participants receiving ergocalciferol 50000 units weekly for 12 weeks
- Ergocalciferol Placebo Group: Participants receiving matching ergocalciferol placebo weekly for 12 weeks
Arm/Group | Ergocalciferol Group | Ergocalciferol Placebo Group
Number analyzed (Participants) | 40 | 50
pg/mL | 74 (42) | 39 (29)
Statistical Analysis 1: Comparison: Ergocalciferol Group; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 12 to 38 weeks
Description: Subjects were monitored during the12 weeks of the intervention at their baseline, week 4, week 8, and week 12 visits for adverse events. Subjects were counseled to contact us after study completion if they had any concerns. During the 26 weeks after study completion, no subject contact the investigative team with an adverse event or concern.
Groups:
- Ergocalciferol Group: Ergocalciferol 50,000 international units once a week for 12 weeks
Arm/Group | Ergocalciferol Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/50
Other Adverse Events (participants affected / at risk) | 0/40 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol Group (N=40) | Placebo Group (N=50)
Asymptomatic hypocalcemia (Endocrine disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes